CLINICAL TRIAL: NCT05770778
Title: Comparison of Inclined Backwalk vs Kneel Walk on Genurecurvatum in Hemiplegic Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sehat Medical Complex (Other)
Responsible Party: Principal Investigator, Waseem Javaid, Project Director, Sehat Medical Complex
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Laraib001-25
Record Dates: First submitted 2023-02-24; First posted 2023-03-15 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-02

CONDITIONS: Hemiplegic Cerebral Palsy
Keywords: Hemiplegic Cerebral Palsy; Genu-Recurvatum; Inclined Backward Walk; Kneel walk.; Treadmill training

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inclined Backward Intervention Group (Active Comparator): Hemiplegic Cerebral Palsy Children
  Interventions: Other: Inclined Backwalk
- Kneel Walk Intervention Group (Active Comparator): Hemiplegic Cerebral Palsy Children
  Interventions: Other: Knee Walk

INTERVENTIONS:
Other: Inclined Backwalk — They will receive inclined backward treadmill gait training exercise for thirty minutes with 2 interval break for 5min every 10 minutes for three times per week over three successive months with a specifically designed physical therapy program according to child need for one hour for each child, three times weekly, over three months.
  Arms: Inclined Backward Intervention Group
Other: Knee Walk — They will receive kneel walk exercise programme for thirty minutes with 2 interval break for 5min every 10 minutes for three times per week over three successive months with a specifically designed physical therapy program according to child need for one hour for each child , three times weekly, over three months.
  Arms: Kneel Walk Intervention Group

SUMMARY:
The 40-68% of ambulating hemiplegic children walk with genu recurvatum and hemiplegic patients shows excessive anterior pelvic tilts (>4 cm) during the stance phase. The objective of the study is to compare the effects of inclined backward treadmill walk vs kneel walk on genu recurvatum in hemiplegic cerebral palsy. 50 participants will be chosen according to inclusion exclusion criteria of the study which will be randomly allocated into two equal groups . One group will receive treadmill training programme with specifically designed physical therapy program according to child need for one hour for each child. And other group will receive kneel walking programme specifically designed physical therapy program according to child need for one hour for each child. The pre and post assessment of genurecurvatum will be assessed by Goniometer.

DETAILED DESCRIPTION:
Efficiency of walking and the development of independent gait are often the focus of therapeutic interventions for children with CP. Motor learning theory suggests that when encountering a new motor skill or adapting a motor skill to a specific situation, a group of interconnected neurons is selected from a primary neuronal repertoire based on prior experience of the task. Generated movement patterns and postural adjustments are then refined via afferent feedback. Therefore, it has been argued that to develop and improve a motor skill such as walking, opportunities for repetitive practice of the skill need to be offered. For this reason use of a mechanical treadmill may improve walking in children with CP. Treadmill walking provides increased opportunity to repetitively train the whole gait cycle, facilitate an improved gait pattern. Improved walking has the potential to increase the mobility and positively influence the societal participation of children with CP at home, at school and in the wider community.

ELIGIBILITY:
Inclusion Criteria:

* GMFM level (I & II)
* knee hyperextension ranged from 10 to 20 degrees

Exclusion Criteria:

* Children with comorbidities (other knee deformities, surgical intervention or fractures) will not included in this study.
* Children who recently have botulinum toxin injection.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-02-03 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Range of Motion | Change from baseline at 3rd Month
  The limit or length ranges of each plane of the joint

CONTACTS AND LOCATIONS:
Overall Officials: Momina Mehmood, Principal Investigator — University of Lahore
Locations (1):
- Sehat Medical Complex, Lahore, Lahore, Punjab Province, Pakistan